CLINICAL TRIAL: NCT06051409
Title: A Pivotal Registrational Phase 3 Study of Olverembatinib Combined With Chemotherapy Versus Imatinib Combined With Chemotherapy in Patients With Newly Diagnosed Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia (Ph+ALL)
Brief Title: A Study of Olverembatinib in Patients With Newly Diagnosed Ph+ALL.
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ascentage Pharma Group Inc. (Industry)
Collaborators: HealthQuest Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HQP1351AG301
Record Dates: First submitted 2023-09-04; First posted 2023-09-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Ph+ ALL
Keywords: Ph+ ALL; Olverembatinib Tablets
MeSH Terms: interventions — olverembatinib; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Olverembatinib (Experimental): Olverembatinib in combination with chemotherapy
  Interventions: Drug: Olverembatinib
- Imatinib (Active Comparator): Imatinib in combination with chemotherapy
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Olverembatinib — Orally, once every other day (QOD).
  Arms: Olverembatinib
Drug: Imatinib — Orally, once daily (QD).
  Arms: Imatinib

SUMMARY:
A global multicenter, open-label, randomized and registrational Phase 3 study to evaluate efficacy and safety of Olverembatinib combined with chemotherapy versus Imatinib combined with chemotherapy in subjects with newly diagnosed Ph+ALL.

DETAILED DESCRIPTION:
Comparing efficacy and safety of Olverembatinib in combination with chemotherapy (investigational arm) vs. Imatinib in combination with chemotherapy (control arm).

ELIGIBILITY:
Inclusion Criteria:

1. Meet the WHO 2016 Ph chromosome or BCR/ABL1 positive Ph+ALL diagnostic and typing criteria for acute lymphoblastic leukemia. This is a newly diagnosed Ph+ALL.
2. Expected survival of at least 3 months.
3. ECOG ≤ 2.
4. Adequate organ function.
5. Use effective contraception during treatment and for at least three months after the last dose of the study drug, and male patients may not donate sperm.
6. Pregnancy test results of serum samples obtained within 7 days prior to the first dosing of a fertile female subject were negative.
7. Understand and voluntarily sign the informed consent approved by the Ethics Committee (EC) and voluntarily complete the study procedure and follow-up examination.

Exclusion Criteria:

1. A history of chronic myeloid leukemia and a diagnosis of acute leukemia with chronic myeloid leukemia.
2. Clinical manifestations of central nervous system (CNS) leukemia or ALL extramedullary infiltration, except lymphadenopathy or hepatosplenomegaly.
3. Previous or current clinical CNS diseases.
4. Autoimmune diseases that may involve the CNS.
5. Use therapeutic doses of anticoagulants and/or antiplatelet agents but allow low doses of anticoagulants to keep central venous lines open.
6. Use a therapeutic drug that has drug interaction with the investigational drug due to other diseases within 7 days prior to the first receipt of the investigational drug.
7. Uncontrolled Heart diseases.
8. Had any VTE in the 6 months prior to randomization, including but not limited to deep vein thrombosis (DVT) or pulmonary embolism.
9. Use of prohibited drugs.
10. The presence of any disease or medical condition that is unstable or may affect its safety or compliance with the study.
11. Medications known to cause prolonged QT interval.
12. Active infections requiring systemic treatment.
13. Disease that severely affects the oral administration and absorption of drugs, or an active gastrointestinal ulcer.
14. Contraindications to the use of glucocorticoids, and the researchers judge that they are not suitable to participate in this study.
15. Bleeding disorders unrelated to the tumor.
16. Plan to undergone major surgery.
17. Allergy to drug ingredients, excipients, or their analogues in the study.
18. Female subjects who are pregnant or breastfeeding or expect to become pregnant during the study plan or within 3 months of the last dosing.
19. Other malignant tumors within 2 years.
20. Any symptom or illness that may interfere with the evaluation of the efficacy and safety of the investigational drug, or any other condition or condition that is not appropriate for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Minimal residual disease negativity rate | Cycles 1 to cycle 3 (each cycle is 28 days)
  The minimal residual disease negativity rate of olverembatinib combined chemotherapy versus imatinib combined chemotherapy in subjects with newly diagnosed Ph+ALL.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0. | Through study completion,an average of 2 years.
  According to CTCAE v5.0, the number and frequency of adverse events of test drug were assessed.
Plasma concentrations of olverembatinib | Cycle 1 to Cycle 3 (each cycle is 28 days)
  Blood samples will be collected to measure the plasma concentration of olverembatinib.
The patients' score of EORTC(The European Organization for Research and Treatment of Cancer) QLQ-C30. | Through study completion,an average of 2 years.
  To evaluate patient-reported outcome in patients treated with olverembatinib plus chemotherapy.（The scale ranges from 0 to 100, with a lower score indicating better quality of life and a higher score on the scale indicating worse symptoms.）

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, M.D.,Ph.D., Principal Investigator — Shanghai Jiaotong University School of Medicine Ruijin Hospital; Suning Chen, M.D.,Ph.D., Principal Investigator — First Affiliated Hospital of Suzhou Medical College
Locations (14):
- Australia (4):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Alfred Health, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Washington
- China (10):
  - The First Affiliated Hospitalo of Bengbu Medical School, Bengbu, Anhui
  - Xinqiao Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Guangdong Province People's Hospital, Guangdong, Guangzhou
  - Nanfang Hospital of Southern Medical University, Guangdong, Guangzhou
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital of Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The first affiliated hospital of Suzhou University, Suzhou, Jiangsu
  - Shanghai Jiao Tong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Institute of blood transfusion of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality